CLINICAL TRIAL: NCT03312387
Title: Cost-effective Strategies to Improve Rehabilitative Outcomes for Heart Failure Patients With Preserved Ejection Fraction
Brief Title: Muscle, Essential Amino Acids, and eXercise in Heart Failure
Acronym: MAAX-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There is no longer any funding to support the study
Sponsor: Arizona State University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jared Dickinson, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00004142
Record Dates: First submitted 2017-10-09; First posted 2017-10-17 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Exercise; Amino Acids, Essential

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essential Amino Acid and Exercise (Experimental): Participants will be provided with essential amino acids during exercise training.
  Interventions: Other: Exercise; Dietary Supplement: Essential Amino Acids
- Placebo and Exercise (Placebo Comparator): Participants will be provided with placebo supplement during exercise training.
  Interventions: Other: Exercise; Dietary Supplement: Placebo

INTERVENTIONS:
Other: Exercise — Aerobic exercise performed 3/d per week during intervention
Dietary Supplement: Essential Amino Acids — Mixture of 10g of essential amino acids ingested throughout intervention
  Arms: Essential Amino Acid and Exercise
Dietary Supplement: Placebo — 10g of maltodextrin ingested throughout intervention
  Arms: Placebo and Exercise

SUMMARY:
Half of heart failure patients have preserved ejection fraction (HFpEF). Like patients with reduced ejection fraction (HFrEF), HFpEF patients suffer from exercise intolerance (low VO2max), which reduces physical function, quality of life, and survival. Strikingly, there is no medication proven to increase survival for HFpEF patients. Whereas exercise intolerance in HFrEF patients is the result of cardiovascular limitations, physical dysfunction in HFpEF patients is largely the result of peripheral abnormalities in skeletal muscle. Indeed, research in HFpEF patients identified that physical function and VO2peak are directly related to leg lean mass, and drugs focused on improving cardiovascular function have failed to improve VO2peak. Unfortunately, no therapy has been identified for this population that can concurrently improve cardiovascular and muscle health. The need for improved muscle therapies is reinforced by the fact that HFpEF patients are commonly older adults who are predisposed to muscle wasting. Strategic essential amino acid (EAA) ingestion has been shown to improve the adaptive response of muscle to exercise. Therefore, the investigators will determine, in HFpEF patients, the extent to which ingesting a strategic mixture of EAAs during an acute aerobic exercise training program enhances the response to this exercise strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+ years of age
* Able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
* Diagnosed with HFpEF as per established echocardiographic criteria (New York Heart Association Class II-III).

Exclusion Criteria:

* Unstable angina, myocardial infarction in the past 4 weeks
* Uncompensated heart failure
* New York Heart Association class IV symptoms, complex ventricular arrhythmias, symptomatic severe aortic stenosis, acute pulmonary embolus, acute myocarditis, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, baseline blood screening abnormalities
* Medication non-compliance
* Medical / orthopedic conditions precluding exercise
* Exercise training (>2 weekly sessions of moderate to high intensity aerobic or resistance exercise)
* Subjects on anti-coagulation medication will not be eligible for the muscle biopsy procedure, but are deemed eligible for study participation if INR < 3.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in VO2max | Change from pre to after the 4 week intervention
  Change in maximal Aerobic Capacity

SECONDARY OUTCOMES:
Change in Flow-mediated Dilation | Change from pre to after the 4 week intervention
  Change in blood vessel function
Change in Pulse wave velocity | Change from pre to after the 4 week intervention
  Change in pulse wave velocity
Change in Diastolic Function | Change from pre to after the 4 week intervention
  Change in diastolic Function
Change in Skeletal Muscle mRNA expression | Change from pre to after the 4 week intervention
  Change in skeletal Muscle mRNA expression

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona State University, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona